CLINICAL TRIAL: NCT00001240
Title: Diagnostic Evaluation of Patients With Suspected Abnormalities of Gastric Secretion
Brief Title: Evaluating Patients With Abnormal Levels of Gastric Acid
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 890005; 89-DK-0005
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-05 (Estimated); Status verified 2004-01

CONDITIONS: Achlorhydria; Gastrinoma; Zollinger Ellison Syndrome
Keywords: Stomach; Hypersecretion; Hyposecretion; Gastrinoma; Zollinger-Ellison Syndrome
MeSH Terms: conditions — Achlorhydria; Gastrinoma; Zollinger-Ellison Syndrome

SUMMARY:
This study is used by the Digestive Diseases Branch to evaluate patients with suspected abnormalities in the secretion of gastric acid. The level of gastric acid is measured by analyzing the gastric juices of each individual patient. The gastric acid sample is obtained by a procedure known as nasogastric suctioning, where a thin plastic tube is passed from the nose to the stomach.

Depending on the patient's present condition further diagnostic testing may be required to achieve a diagnosis.

DETAILED DESCRIPTION:
This study is an omnibus protocol used by the Digestive Diseases Branch to evaluate patients with suspected abnormalities of gastric acid secretion. Gastric acid secretion is measured by means of analysis of gastric juices obtained by nasogastric suction. Other clinically indicated diagnostic procedures are performed depending on the patient's clinical state in order to reach a diagnosis.

ELIGIBILITY:
Eligibility criteria not identified in the protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1989-01; Study Completion 2004-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK), Bethesda, Maryland, United States

REFERENCES:
- [Background] McArthur KE, Collen MJ, Maton PN, Cherner JA, Howard JM, Ciarleglio CA, Cornelius MJ, Jensen RT, Gardner JD. Omeprazole: effective, convenient therapy for Zollinger-Ellison syndrome. Gastroenterology. 1985 Apr;88(4):939-44. doi: 10.1016/s0016-5085(85)80011-1. PMID 3972233
- [Background] Howard JM, Chremos AN, Collen MJ, McArthur KE, Cherner JA, Maton PN, Ciarleglio CA, Cornelius MJ, Gardner JD, Jensen RT. Famotidine, a new, potent, long-acting histamine H2-receptor antagonist: comparison with cimetidine and ranitidine in the treatment of Zollinger-Ellison syndrome. Gastroenterology. 1985 Apr;88(4):1026-33. doi: 10.1016/s0016-5085(85)80024-x. PMID 2857672
- [Background] Vinayek R, Howard JM, Maton PN, Wank SA, Slaff JI, Gardner JD, Jensen RT. Famotidine in the therapy of gastric hypersecretory states. Am J Med. 1986 Oct 24;81(4B):49-59. doi: 10.1016/0002-9343(86)90600-5. PMID 2877575